CLINICAL TRIAL: NCT06508996
Title: Clinical Evaluation of the Xpert® HCV Test on the GeneXpert® Xpress System
Brief Title: Xpert Hepatitis-C Virus (HCV) Test on the GeneXpert Xpress System
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: 293C
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: HCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — capillary and venous whole blood collected from consented individuals with signs and symptoms and/or individuals at-risk of HCV infection, irrespective of HCV antibody status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Capillary whole blood: Capillary whole blood from individuals with signs and symptoms and/or at-risk of HCV infection
  Interventions: Diagnostic Test: Xpert HCV

INTERVENTIONS:
Diagnostic Test: Xpert HCV — Detection of HCV RNA by Xpert HCV test

SUMMARY:
A multi-site prospective, all comers study that was conducted at geographically diverse locations in the United States.

DETAILED DESCRIPTION:
Whole blood specimens were collected from consented individuals with signs and symptoms and/or individuals at-risk of HCV infection, irrespective of HCV antibody status at a single timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Participant was ≥18 years old
* Participant was not on treatment at time of enrollment based on review of medical records or self-reported
* Participant had signs and symptoms and/or is considered at-risk of HCV infection

Exclusion Criteria:

* Clinician assessed that the participant was not suitable for inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Specimens collected from individuals showing signs and symptoms and/or at risk of HCV infection
Sampling Method: Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Percent Agreement compared to Patient infected status (PIS) | 1 day
  Clinical performance comparing Xpert test to PIS (NAAT + Antibody status)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Havens, Principal Investigator — University of Kentucky College of Medicine
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No